CLINICAL TRIAL: NCT02140047
Title: Exploratory Clinical Study of MT-2301 in Healthy Infants (Phase 2)
Brief Title: Exploratory Clinical Study of MT-2301
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MT-2301-J01
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Haemophilus Influenza Type b
Keywords: Haemophilus influenza type b; Hib
MeSH Terms: conditions — Haemophilus Infections | interventions — Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MT-2301-Low (Experimental)
  Interventions: Biological: Haemophilus b conjugate vaccine diphteria CRM197 protein conjugate)-Low + DPT-IPV
- MT-2301-High (Experimental)
  Interventions: Biological: Haemophilus b conjugate vaccine diphteria CRM197 protein conjugate)-High + DPT-IPV
- ActHIB (Active Comparator)
  Interventions: Biological: Haemophilus influenza type b conjugate vaccine + DPT-IPV

INTERVENTIONS:
Biological: Haemophilus b conjugate vaccine diphteria CRM197 protein conjugate)-Low + DPT-IPV — 0.25mL, subcutaneous injection
  Other Names: MT-2301-Low + Tetrabik®
  Arms: MT-2301-Low
Biological: Haemophilus b conjugate vaccine diphteria CRM197 protein conjugate)-High + DPT-IPV — 0.5mL, subcutaneous injection
  Other Names: MT-2301-High + Tetrabik®
  Arms: MT-2301-High
Biological: Haemophilus influenza type b conjugate vaccine + DPT-IPV — 0.5mL, subcutaneous injection
  Other Names: ActHIB® + Tetrabik®
  Arms: ActHIB

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of MT-2301 when co-administered with DPT-IPV using ActHIB® as a control in healthy infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged ≥2 and <7 months at the first vaccination of the study drug
* Written informed consent is obtained from a legal guardian (parent)

Exclusion Criteria:

* With obvious pyrexia (axillary temperature of 37.5ºC or higher) at vaccination of the study drug
* With known serious acute disease
* With known underlying disease such as cardiovascular disease, renal disease, hepatic disease, blood dyscrasia, and respiratory disease
* With past diagnosis of immunodeficiency or currently under immunosuppressive treatment
* History of anaphylaxis due to food or pharmaceuticals
* With experience of Hib infection, diphtheria, pertussis, tetanus, and acute poliomyelitis
* With experience of Hib vaccination, or administration of vaccine including either diphtheria, pertussis, tetanus, or polio as a constituent
* History of convulsions
* Administered a live vaccine within 27 days before the first vaccination of the study drug, or inactivated vaccine or toxoid within 6 days before vaccination
* Administered transfusion, immunosuppressant (excluding drugs for external use), or immunoglobulin formulation
* Administered corticosteroid 2 mg/kg per day or more as prednisolone (excluding drugs for external use) continuously for more than 1 week
* Participated in other studies within 12 weeks before obtaining consent

Ages: 2 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Nakano, M.D., Ph.D., Study Director — Department of pediatrics, Kawasaki Hospital, Kawasaki Medical School
Locations (1):
- Investigational site, Fukuoka, Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- MT-2301-Low: Haemophilus b conjugate vaccine diphteria CRM197 protein conjugate-Low
- MT-2301-High: Haemophilus b conjugate vaccine diphteria CRM197 protein conjugate-High
- ActHIB: Haemophilus influenza type b conjugate vaccine
Period: Overall Study
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Started | 52 | 52 | 50
Completed | 51 | 51 | 50
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by parent/guardian | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB | Total
Number analyzed (Participants) | 52 | 52 | 50 | 154
Age, Customized [Count of Participants; unit: Participants]
  >=2 and <3 months | 43 | 39 | 37 | 119
  >=3 months | 9 | 13 | 13 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 20 | 64
  Male | 29 | 31 | 30 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Japanese) | 52 | 52 | 50 | 154

OUTCOME MEASURES:

1. Primary Outcome: Antibody Prevalence Rate Against Anti-PRP With 1 μg/mL or Higher, Defined as the Percentage of Participants With the Antibody Against Anti-PRP
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects 154.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Number analyzed (Participants) | 52 | 52 | 50
percentage of participants | 100.0 [93.2 to 100.0] | 96.2 [86.8 to 99.5] | 94.0 [83.5 to 98.7]

2. Secondary Outcome: Anti-PRP Antibody Prevalence Rate With 0.15 μg/mL or Higher, Defined as the Percentage of Participants With the Anti-PRP Antibody
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects 154.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Number analyzed (Participants) | 52 | 52 | 50
percentage of participants | 100.0 [93.2 to 100.0] | 100.0 [93.2 to 100.0] | 100.0 [92.9 to 100.0]

3. Secondary Outcome: Geometric Mean Antibody Titer of Anti-PRP Antibody
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects 154.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Number analyzed (Participants) | 52 | 52 | 50
µg/mL | 21.120 [16.233 to 27.495] | 13.724 [10.077 to 18.690] | 7.374 [5.212 to 10.434]

4. Secondary Outcome: Anti-PRP Antibody Prevalence Rate With 1 μg/mL or Higher, Defined as the Percentage of Participants With the Anti-PRP Antibody
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: For antibody analysis at Visit 6, number of subjects decreased from 154 to 152.MT-2301-Low group: due to withdrawal by parent/guardian (n=1) . MT-2301-High group: due to withdrawal by parent/guardian (n=1) .
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Number analyzed (Participants) | 51 | 51 | 50
percentage of participants | 100.0 [93.0 to 100.0] | 100.0 [93.0 to 100.0] | 100.0 [92.9 to 100.0]

5. Secondary Outcome: Anti-PRP Antibody Prevalence Rate With 0.15 μg/mL or Higher, Defined as the Percentage of Participants With the Anti-PRP Antibody
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Number analyzed (Participants) | 51 | 51 | 50
percentage of participants | 100.0 [93.0 to 100.0] | 100.0 [93.0 to 100.0] | 100.0 [92.9 to 100.0]

6. Secondary Outcome: Geometric Mean Antibody Titer of Anti-PRP Antibody
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Number analyzed (Participants) | 51 | 51 | 50
µg/mL | 65.086 [52.241 to 81.089] | 48.448 [35.066 to 66.936] | 39.752 [29.379 to 53.787]

7. Secondary Outcome: Geometric Mean Antibody Titer Against Diphtheria Toxin
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects 154. MT-2301-High group number of subjects further decreased due to insufficient sample volume (diphtheria :n=1)
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Number analyzed (Participants) | 52 | 51 | 50
IU/mL | 1.026 [0.746 to 1.410] | 1.016 [0.777 to 1.329] | 1.110 [0.824 to 1.497]

8. Secondary Outcome: Geometric Mean Antibody Titer Against Pertussis
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects 154.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Number analyzed (Participants) | 52 | 52 | 50
U/mL
  pertussis （PT） | 189.03 [162.60 to 219.77] | 191.62 [168.87 to 217.43] | 203.58 [181.78 to 227.98]
  pertussis （FHA） | 54.82 [47.23 to 63.62] | 44.50 [37.24 to 53.18] | 68.75 [57.37 to 82.37]

9. Secondary Outcome: Geometric Mean Antibody Titer Against Tetanus Toxin
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects 154.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Number analyzed (Participants) | 52 | 52 | 50
U/mL | 0.575 [0.449 to 0.738] | 0.497 [0.374 to 0.660] | 0.542 [0.373 to 0.786]

10. Secondary Outcome: Fold Change in Geometric Mean Antibody Titer Against Polio Virus
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects 154. MT-2301-High group number of subjects further decreased due to insufficient sample volume (polio serotype1,2 and 3: n=3 each) . MT-2301-Low group number of subjects further decreased due to insufficient sample volume (polio serotype1,2 and 3: n=2 each). ActHIV group number of subjects further decreased due to insufficient sample volume (polio serotype1,2 and 3: n=1 each).
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Number analyzed (Participants) | 50 | 49 | 49
fold change
  polio virus serotype 1 | 1468.4 [1017.4 to 2119.2] | 1554.3 [1094.5 to 2207.3] | 1790.5 [1192.6 to 2688.0]
  polio virus serotype 2 | 2272.4 [1809.2 to 2854.2] | 2776.0 [2266.4 to 3400.2] | 2896.3 [2311.9 to 3628.4]
  polio virus serotype 3 | 2574.4 [2061.6 to 3214.7] | 1976.8 [1569.1 to 2490.6] | 2198.1 [1699.9 to 2842.3]

11. Secondary Outcome: Geometric Mean Antibody Titer Against Diphtheria Toxin
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: For antibody analysis at Visit 6, number of subjects 152.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Number analyzed (Participants) | 51 | 51 | 50
IU/mL | 9.831 [7.856 to 12.302] | 10.102 [8.195 to 12.454] | 9.511 [7.616 to 11.876]

12. Secondary Outcome: Geometric Mean Antibody Titer Against Pertussis
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: For antibody analysis at Visit 6, number of subjects 152.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Number analyzed (Participants) | 51 | 51 | 50
U/mL
  pertussis （PT） | 239.48 [200.45 to 286.11] | 233.12 [200.58 to 270.94] | 262.73 [223.61 to 308.69]
  pertussis （FHA） | 124.84 [104.61 to 148.99] | 119.41 [98.56 to 144.68] | 158.85 [126.24 to 199.89]

13. Secondary Outcome: Geometric Mean Antibody Titer Against Tetanus Toxin
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: For antibody analysis at Visit 6, number of subjects 152.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Number analyzed (Participants) | 51 | 51 | 50
U/mL | 1.750 [1.412 to 2.169] | 1.726 [1.374 to 2.169] | 2.051 [1.429 to 2.943]

14. Secondary Outcome: Fold Change in Geometric Mean Antibody Titer Against Polio Virus
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: For antibody analysis at Visit 6, number of subjects 152. MT-2301-High group number of subjects further decreased due to insufficient sample volume (polio serotype1: n=1) . ActHIV group number of subjects further decreased due to insufficient sample volume (polio serotype1,2 and 3: n=1 each).
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
Number analyzed (Participants) | 51 | 51 | 50
fold change
  polio virus serotype 1: number analyzed (Participants) | 51 | 50 | 49
  polio virus serotype 1 | 3479.6 [2487.6 to 4867.2] | 4544.8 [3303.0 to 6253.5] | 4685.1 [3194.4 to 6873.7]
  polio virus serotype 2: number analyzed (Participants) | 51 | 51 | 49
  polio virus serotype 2 | 8360.7 [6703.5 to 10427.7] | 9908.9 [8030.0 to 12227.5] | 10642.5 [8809.5 to 12856.9]
  polio virus serotype 3: number analyzed (Participants) | 51 | 51 | 49
  polio virus serotype 3 | 6681.2 [5410.1 to 8250.9] | 7448.6 [5811.4 to 9546.9] | 7578.8 [5756.2 to 9978.6]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year
Arm/Group | MT-2301-Low | MT-2301-High | ActHIB
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52 | 0/50
Serious Adverse Events (participants affected / at risk) | 4/52 | 2/52 | 2/50
Other Adverse Events (participants affected / at risk) | 52/52 | 52/52 | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-2301-Low (N=52) | MT-2301-High (N=52) | ActHIB (N=50)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MT-2301-Low (N=52) | MT-2301-High (N=52) | ActHIB (N=50)
Eye discharge (Eye disorders) | 3 | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 3 | 6
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 5
Crying (General disorders) | 13 | 13 | 16
Injection site bruising (General disorders) | 3 | 0 | 0
Injection site erythema (General disorders) | 39 | 41 | 36
Injection site induration (General disorders) | 34 | 30 | 22
Injection site pain (General disorders) | 8 | 9 | 8
Injection site swelling (General disorders) | 26 | 21 | 17
Irritability postvaccinal (General disorders) | 19 | 24 | 22
Pyrexia (General disorders) | 40 | 36 | 41
Bronchitis (Infections and infestations) | 7 | 4 | 4
Conjunctivitis (Infections and infestations) | 8 | 5 | 3
Exanthema subitum (Infections and infestations) | 6 | 3 | 5
Gastroenteritis (Infections and infestations) | 5 | 6 | 2
Hand-foot-and-mouth disease (Infections and infestations) | 6 | 3 | 5
Herpangina (Infections and infestations) | 3 | 1 | 1
Nasopharyngitis (Infections and infestations) | 14 | 17 | 9
Otitis media (Infections and infestations) | 5 | 5 | 4
Pharyngitis (Infections and infestations) | 4 | 2 | 1
Respiratory syncytial virus infection (Infections and infestations) | 2 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 4
Arthropod sting (Injury, poisoning and procedural complications) | 6 | 5 | 3
Decreased appetite (Metabolism and nutrition disorders) | 9 | 11 | 12
Hypersomnia (Nervous system disorders) | 19 | 21 | 11
Insomnia (Psychiatric disorders) | 11 | 13 | 18
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 16 | 20 | 14
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 7 | 9 | 2
Eczema (Skin and subcutaneous tissue disorders) | 11 | 5 | 8
Eczema infantile (Skin and subcutaneous tissue disorders) | 3 | 3 | 5
Miliaria (Skin and subcutaneous tissue disorders) | 8 | 7 | 5
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other